CLINICAL TRIAL: NCT06582797
Title: Analytical Treatment Interruption in a Patient With HIV Post Allogeneic Stem Cell Transplantation From a CCR5 delta32 Homozygous Donor
Acronym: ATI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Wissam El Atrouni, Associate Professor, University of Kansas Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 160833
Record Dates: First submitted 2024-08-30; First posted 2024-09-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: HIV-1-infection
Keywords: stem cell transplant; HIV proof of cure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment withdraw (Experimental): patient with discontinue standard of care treatment for their HIV infection
  Interventions: Other: discontinuation of ART

INTERVENTIONS:
Other: discontinuation of ART — patient will discontinue their standard of care HIV treatment with ART while being closely monitored

SUMMARY:
Patients who have Human Immunodeficiency Virus-1 (HIV-1) infection, who also had a stem cell transplant may have achieved cure of their HIV infection. Once the patients blood shows no detectable levels of HIV virus in their blood collected from a process called leukapheresis, they will be closely monitored while discontinuing their HIV treatment which is know as antiretroviral therapy or, ART. They will be tested regularly and monitored for up to 52 weeks at which point they may be considered cured of their HIV.

DETAILED DESCRIPTION:
On week -1, a HIV VL and CD4 count will be drawn. If VL remains undetectable, at study week 0, and no other exclusion criteria noted, subject will discontinue ART and enter ATI phase of the study. HIV-1 plasma VL will be monitored every 2 weeks for 52 weeks, then patient returns under the care of their HIV provider. CD4 T cell count will be monitored every 4 weeks.

Depressions symptom check with PHQ-9 check monthly with study visits. Since patients might be cured and at risk of acquiring HIV during the period of treatment interruption, they will be offered Prep on Demand (Truvada) to be used no more than once a month (with notification of study PI when it happens). When Prep on Demand is used, we will ask patient to come in for ART drug level measurement same week.

If patient meets any of the restart ART criteria during the interruption phase, they will discontinue the ATI phase of study and re-start ART and enter the follow up ART phase. If subject maintains undetectable plasma HIV VL (assay quantification threshold 20 copies/mL), they will remain off ART and continue to be monitored until restart criteria are met. If patient meets the restart criteria, they will be followed for 12 months post re-initiation of therapy by their HIV provider. The first month post restart of therapy will require weekly visits, followed by monthly visits thereafter until HIV VL is back <50 copies/mL. Leukapheresis (per previously approved protocol that patient consented to) will be performed at 6 months and 12 months post ATI if in continued viral remission.

ELIGIBILITY:
Inclusion Criteria:

* Positive HIV testing
* Has undergone a stem cell transplant

Exclusion Criteria:

* under 18 years of age
* unwilling to comply with protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2034-09 (Estimated); Study Completion 2034-09 (Estimated)

PRIMARY OUTCOMES:
Proof of cure | 52 weeks
  patient will prove cured of HIV infection if no viral load tests result positive over the duration of study

IPD SHARING:
Plan to Share IPD: No